CLINICAL TRIAL: NCT04202146
Title: Cannabis Use and Relapse After One Week of Contingency Management Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000023188
Record Dates: First submitted 2019-01-09; First posted 2019-12-17 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Cannabis Dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contingency Management + Motivational Interviewing (Experimental): Participants will complete a seven-day combined CM with two sessions of brief Motivation Interviewing (MI) followed by standardized individual drug counseling.
  Interventions: Behavioral: Contingency Management + Motivational Interviewing

INTERVENTIONS:
Behavioral: Contingency Management + Motivational Interviewing — Seven-day combined CM with two sessions of brief Motivation Interviewing (MI) followed by standardized individual drug counseling on cannabis use and relapse.

SUMMARY:
The purpose of this study is to examine the effects of a seven-day combined contingency management (CM) with two sessions of brief Motivation Interviewing (MI) followed by standardized individual drug counseling on cannabis use and relapse in the following 90-day period in individuals with moderate to severe Cannabis Use Disorder (DSM-5).

DETAILED DESCRIPTION:
The primary aim of this study is to examine cannabis use and rates of abstinence and relapse in individuals with moderate to severe Cannabis Use Disorder (CUD) after intensive 7-day contingency management (CM) procedure to reinforce abstinence from cannabis use. In addition, this study will evaluate the effect of CM with two sessions of brief MI on the severity of cannabis withdrawal signs during the first 7-days of CM treatment and then during the following month.

The study will also focus on prospectively monitoring the sustenance of abstinence and time to lapse and relapse to cannabis use over a 90-day period, using ecological momentary assessment (EMA) via a smartphone-based application. An additional aim will be to evaluate changes in symptoms of CUD during the period following the 7-day using the diagnostic criteria of the DSM-5.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) less than 32;
* Good health as verified by screening examination;
* Able to read English and complete study evaluations;
* Able to provide informed written and verbal consent;
* CUD sample must meet DSM-5 criteria for CUD as assessed using SCID-I and have positive cannabis urine toxicology screens on admission to study, with weekly 3 or more days of self-reported cannabis use.

Exclusion Criteria:

* Meet current DSM-5 criteria for dependence on another psychoactive substance or alcohol, excluding nicotine and mild Alcohol Use Disorder
* Current use of opiates or history of opiate abuse/dependence;
* Regular use of anticonvulsants, sedatives/hypnotics, prescription analgesics, other antihypertensives, anti-arrythmics, antiretroviral medications, tricyclic antidepressants, SSRI's, naltrexone, antabuse;
* Psychotic or otherwise severely psychiatrically disabled (i.e., suicidal, homicidal, current mania);
* Significant underlying medical conditions such as a history of seizure disorder, cerebral, renal, thyroid or cardiac pathology which in the opinion of study physician would preclude subjects from fully cooperating or be of potential harm during the study; a known history of Hepatitis B, C, or HIV infection;
* Any psychotic disorder or current Axis I psychiatric symptoms (excluding anxiety disorders) requiring specific attention, including need for psychiatric medications
* Women who are pregnant, nursing or refuse to use a reliable form of birth control (as assessed by pregnancy urine test during initial intake appointment; and
* Traumatic brain injury or extended loss of consciousness.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Cannabis Use | Slope Change 12 Weeks
  The Structured Clinical Interview for DSM-V (SCID-II) will be used to ascertain DSM-5 Axis 1 psychiatric and substance abuse diagnoses (First, et al., 2015) and specifically to determine presence/absence of DSM-5 Cannabis Use Disorder (CUD). The SCID-II interview for cannabis use will be administered at intake and weeks 4, 8, and 12 to measure changes in problematic cannabis use. The outcome will be the slope of change over study day in daily quantity of use and the percent use days per week. In addition, we will measure the percent of individuals who experienced a relapse throughout the study by week 12 (3 days of use weekly or 3 consecutive days of use).
Overall Drug Use | Slope Change 12 Weeks
  The Time-Line Follow-Back Interview will also be used to assess cannabis, alcohol, other drugs and nicotine use in the previous ninety days, during the study and during follow-up. This is a reliable experimenter-administered assessment (Sobell and Sobell, 1992), which uses a calendar prompt to facilitate recall of drug use during a targeted period, and well-validated in alcohol and drug abuse treatment studies (Fals-Stewart et al., 2000). This questionnaire will be administered at intake and weekly. The outcome will be the slope of change over study day in daily quantity of use and the percent use days per week. In addition, we will measure the percent of individuals who experienced a relapse throughout the study by week 12 (3 days of use weekly or 3 consecutive days of use).
Cannabis Use Severity | Slope Change 12 Weeks
  The Cannabis Use Disorder Identification Test-Revised (CUDIT) is an 8-item scale that will be used to quantify the severity of cannabis use over the past six-months (Adamson et al., 2010). This questionnaire will be administered at intake and weeks 4, 8, and 12. A summed score is used as an outcome where higher equals more cannabis-related problems.
Urine Toxicology for Quantitative THC levels | Slope Change 12 Weeks
  A urine drug screen will be given at each visit during week 1 to reinforce using CM for cannabis abstinence and monitor progressive reduction in THC levels, and at each visit during the duration of the study to assess levels of THC for determination of the primary clinical outcome of cannabis relapse. The slope of change over weeks 1 through 12 in quantitative THC levels and metabolites will be the outcome measure.
Urine Toxicology for Quantitative THC metabolites | Slope Change 12 Weeks
  A urine drug screen will be given at each visit during week 1 to reinforce using CM for cannabis abstinence and monitor progressive reduction in THC levels, and at each visit during the duration of the study to assess levels of THC for determination of the primary clinical outcome of cannabis relapse. The slope of change over weeks 1 through 12 in quantitative THC levels and metabolites will be the outcome measure.

SECONDARY OUTCOMES:
Cannabis Withdrawal | Slope Change 12 Weeks
  The Cannabis Withdrawal Scale (Allsop et al., 2011):Participants will complete this questionnaire during weekly visits and during the EMA evening survey. The 19-item CWS has excellent reliability and has been validated in several previous cannabis abstinence, self-administration and treatment studies (Budney et al., 1999; Budney & Moore, 2002; Haney, 2002). Participants will indicate if they experienced these symptoms, the degree to which they experienced them (0=Not at all to 10=Extremely), and how much of an impact it had on their lives (0=No at all to 10=Extremely). A summed scores, where a higher score means more difficulty, will be used as the outcome. The slope of change in the number of symptoms endorsed weekly will be the secondary outcome measure.

OTHER OUTCOMES:
Marijuana Intoxication | Baseline and Week 1
  The Marijuana Intoxication Assessment will be used to assess acute cannabis intoxication at each visit using a brief structured interview conducted by the trained research staff member. This 8-item will be measured at intake and during the first week. This is a screen to ensure compliance with study requirements.

CONTACTS AND LOCATIONS:
Locations (1):
- The Yale Stress Center: Yale University, New Haven, Connecticut, United States